CLINICAL TRIAL: NCT01204749
Title: A Phase 3, Randomized, Double-Blind Trial of Weekly Paclitaxel Plus AMG 386 or Placebo in Women With Recurrent Partially Platinum Sensitive or Resistant Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancers
Brief Title: TRINOVA-1: A Study of AMG 386 or Placebo, in Combination With Weekly Paclitaxel Chemotherapy, as Treatment for Ovarian Cancer, Primary Peritoneal Cancer and Fallopian Tube Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20090508
Record Dates: First submitted 2010-08-26; First posted 2010-09-17 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cancer
Keywords: AMGEN; AMG 386; Angiogenesis Inhibitors; Fallopian Tube Cancer; Primary Peritoneal Cancer; Paclitaxel; Ovarian Cancer; TRINOVA-1
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — trebananib; Angiogenesis Inhibitors; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMG 386 (Experimental): Arm A: Paclitaxel 80mg/m2 IV QW and Blinded AMG 386 15mg/kg IV QW
  Interventions: Drug: AMG 386; Drug: Paclitaxel
- AMG 386 Placebo (Placebo Comparator): Arm B: Paclitaxel 80mg/m2 IV QW and Blinded AMG 386 Placebo IV QW
  Interventions: Drug: AMG 386 Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: AMG 386 — Weekly Intravenous (IV) AMG 386 15 mg/kg
  Other Names: Angiogenesis inhibitor
  Arms: AMG 386
Drug: AMG 386 Placebo — Weekly Intravenous (IV) placebo 15 mg/kg
  Other Names: Placebo comparator
  Arms: AMG 386 Placebo
Drug: Paclitaxel — Paclitaxel 80 mg/m2 intravenous (IV) weekly (3 on/1 off)
  Other Names: Taxol USPI, 2007; Taxol SPC, 2009
  Arms: AMG 386
Drug: Paclitaxel — Paclitaxel 80 mg/m2 intravenous (IV) weekly (3 on/1 off)
  Other Names: Taxol USPI, 2007; Taxol SPC, 2009
  Arms: AMG 386 Placebo

SUMMARY:
The purpose of this study is to determine if treatment with paclitaxel plus AMG 386 is superior to paclitaxel plus placebo in women with recurrent partially platinum sensitive or resistant epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer.

AMG 386 is a man-made medication that is designed to stop the development of blood vessels in cancer tissues. Cancer tissues rely on the development of new blood vessels, a process called angiogenesis, to obtain a supply of oxygen and nutrients to grow.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age or older at the time the written informed consent is obtained
* Gynecologic Oncology Group (GOG) Performance Status of 0 or 1
* Life expectancy >= 3 months (per investigator opinion)
* Histologically or cytologically documented invasive epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer (Subjects with pseudomyxoma , mesothelioma, unknown primary tumor, sarcoma, or neuroendocrine histology, with borderline ovarian cancer, ie, subjects with low malignant potential tumors, and with clear cell or mucinous histology are excluded)
* Subjects must have undergone surgery for ovarian cancer, primary peritoneal cancer, or fallopian tube cancer including at least a unilateral oophorectomy
* Radiologically evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 with modifications
* Subjects must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation therapy, bevacizumab or extended therapy administered after surgical or non-surgical assessment.
* Adequate organ and hematological function
* Generally well controlled blood pressure with systolic blood pressure <= 140 mmHg and diastolic blood pressure <= 90 mmHg prior to randomization. The use of anti-hypertensive medications to control hypertension is permitted
* Radiographically documented disease progression either on or following the last dose of prior chemotherapy regimen for epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer

Exclusion Criteria:

* Subjects who have received more than 3 previous regimens of anti-cancer therapy for epithelial ovarian, primary peritoneal or fallopian tube cancers
* Subjects who have received paclitaxel as consolidation therapy, maintenance, or monotherapy are excluded
* Subjects with primary platinum-refractory disease
* Subjects with platinum-free interval (PFI) > 12 months from their last platinum based therapy
* Radiotherapy <= 14 days prior to randomization. Subjects must have recovered from all radiotherapy-related toxicities
* Previous abdominal or pelvic radiotherapy
* History of arterial or venous thromboembolism within 12 months prior to randomization
* History of clinically significant bleeding within 6 months prior to randomization
* History of central nervous system metastasis
* Has not yet completed a 21 day washout period prior to randomization for any previous anti cancer systemic therapies (30 days for prior bevacizumab)
* Enrolled in or has not yet completed at least 30 days (prior to randomization) since ending other investigational device or drug, or currently receiving other investigational treatments
* Unresolved toxicities from prior systemic therapy that are Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 >= Grade 2 in severity except alopecia
* Known active or ongoing infection (except uncomplicated urinary tract infection [UTI]) within 14 days prior to randomization
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Treatment within 30 days prior to randomization with strong immune modulators including but not limited to systemic cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, thalidomide, and lenalidomide
* Clinically significant cardiovascular disease within 12 months prior to randomization
* Major surgery within 28 days prior to randomization or still recovering from prior surgery
* Minor surgical procedures, except placement of tunneled central venous access device within 3 days prior to randomization. Diagnostic laparoscopy is regarded as a minor surgical procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 8 Months on average

SECONDARY OUTCOMES:
Overall survival | 20 months on average
Objective Response Rate | From Baseline (if subject has Measurable Disease) until objective response (radiologic)
Duration of response | From Baseline until progression
CA-125 response rate per Gynecologic Cancer Intergroup (GCIG) and change in CA-125 | From Baseline until CA-125 response
Incidence of adverse events and significant laboratory abnormalities | 8 Months on average
Pharmacokinetics of AMG 386 (Cmax and Cmin) | Week 1 until week 9 of treatment
Incidence of the occurrence of anti-AMG 386 antibody formation | Week 1 until maximum of 1-year following last dose of study drug
Patient reported Health Related Quality of Life (HRQOL) and ovarian cancer related symptoms using Functional Assessment of Cancer Therapy - Ovary questionnaire (FACT-O) | From week 1 until 30-days following last study drug administration
Overall health status using EuroQOL(EQ-5D) | From week 1 until 30-days following last study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (193):
- United States (29):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Stanford, California
  - Research Site, Englewood, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Hollywood, Florida
  - Research Site, Orlando, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Peoria, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Metairie, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, Hackensack, New Jersey
  - Research Site, Brightwaters, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Abington, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (7):
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Greenslopes, Queensland
  - Research Site, Bendigo, Victoria
  - Research Site, Bentleigh East, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Parkville, Victoria
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Namur
- Brazil (5):
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, ItajaÃ-, Santa Catarina
  - Research Site, Ribeirão Preto, SÃ£o Paulo
  - Research Site, SÃ£o Paulo, SÃ£o Paulo
- Bulgaria (5):
  - Research Site, Gabrovo
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Chile (2):
  - Research Site, Temuco, CautÃ-n
  - Research Site, Valparaíso, ValparaÃ-so
- Research Site, Zagreb, Croatia
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (24):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, OrlÃ©ans Cedex 2
  - Research Site, Paris
  - Research Site, PÃ©rigueux Cedex
  - Research Site, Reims
  - Research Site, Saint GrÃ©goire Cedex
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Villejuif
- Greece (5):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- India (4):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
- Israel (5):
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Kefar Sava
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (9):
  - Research Site, Benevento
  - Research Site, Catania
  - Research Site, Cosenza (CS)
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Potenza
  - Research Site, Roma
- Japan (14):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kure, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Morioka, Iwate
  - Research Site, Niigata, Niigata
  - Research Site, Sayama, Osaka
  - Research Site, Hidaka-Shi, Saitama
  - Research Site, Suntou-gun, Shizuoka
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Yonago, Tottori
  - Research Site, Kurume
  - Research Site, Tokyo
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Malaysia (3):
  - Research Site, Johor Bahru, Johor
  - Research Site, Kota Bharu, Kelantan
  - Research Site, Kuala Lumpur, Kuala Lumpur
- Mexico (3):
  - Research Site, Distrito Federal, Mexico City
  - Research Site, Mexico City, Mexico City
  - Research Site, San Luis Potosí City, San Luis PotosÃ-
- Research Site, Lima, Lima Province, Peru
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (5):
  - Research Site, Coimbra
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Santa Maria da Feira
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Suceava
  - Research Site, Târgu Mureş
- Russia (8):
  - Research Site, Ivanovo
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Voronezh
- Research Site, Ljubljana, Slovenia
- South Africa (6):
  - Research Site, Groenkloof, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Kraaifontein, Western Cape
  - Research Site, Observatory
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seoul
- Spain (14):
  - Research Site, CÃ³rdoba, AndalucÃ-a
  - Research Site, Huelva, AndalucÃ-a
  - Research Site, MÃ¡laga, AndalucÃ-a
  - Research Site, Seville, AndalucÃ-a
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Salamanca, Castilla LeÃ³n
  - Research Site, Badalona, CataluÃ±a
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Vigo, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, San SebastiÃ¡n, PaÃ-s Vasco
  - Research Site, Elche, Valencia
  - Research Site, Valencia, Valencia
- Sweden (2):
  - Research Site, UmeÃ¥
  - Research Site, Uppsala
- Switzerland (5):
  - Research Site, Baden
  - Research Site, Bellinzona
  - Research Site, Chur
  - Research Site, Geneva
  - Research Site, Zurich
- United Kingdom (6):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Nottingham
  - Research Site, Poole
  - Research Site, Sutton

REFERENCES:
- [Background] Monk BJ, Poveda A, Vergote I, Raspagliesi F, Fujiwara K, Bae DS, Oaknin A, Ray-Coquard I, Provencher DM, Karlan BY, Lhomme C, Richardson G, Rincon DG, Coleman RL, Herzog TJ, Marth C, Brize A, Fabbro M, Redondo A, Bamias A, Tassoudji M, Navale L, Warner DJ, Oza AM. Anti-angiopoietin therapy with trebananib for recurrent ovarian cancer (TRINOVA-1): a randomised, multicentre, double-blind, placebo-controlled phase 3 trial. Lancet Oncol. 2014 Jul;15(8):799-808. doi: 10.1016/S1470-2045(14)70244-X. Epub 2014 Jun 17. PMID 24950985
- [Background] Monk BJ, Poveda A, Vergote I, Raspagliesi F, Fujiwara K, Bae DS, Oaknin A, Ray-Coquard I, Provencher DM, Karlan BY, Lhomme C, Richardson G, Rincon DG, Coleman RL, Marth C, Brize A, Fabbro M, Redondo A, Bamias A, Ma H, Vogl FD, Bach BA, Oza AM. Final results of a phase 3 study of trebananib plus weekly paclitaxel in recurrent ovarian cancer (TRINOVA-1): Long-term survival, impact of ascites, and progression-free survival-2. Gynecol Oncol. 2016 Oct;143(1):27-34. doi: 10.1016/j.ygyno.2016.07.112. Epub 2016 Aug 18. PMID 27546885
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Fujiwara K, Monk BJ, Lhomme C, Coleman RL, Brize A, Oaknin A, Ray-Coquard I, Fabbro M, Provencher D, Bamias A, Vergote I, DeCensi A, Zhang K, Vogl FD, Bach BA, Raspagliesi F. Health-related quality of life in women with recurrent ovarian cancer receiving paclitaxel plus trebananib or placebo (TRINOVA-1). Ann Oncol. 2016 Jun;27(6):1006-1013. doi: 10.1093/annonc/mdw147. Epub 2016 Mar 30. PMID 27029706
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com